CLINICAL TRIAL: NCT04471805
Title: Estrogen Levels and Leg Muscle Fatigability in Eumenorrheic Young Women After 4 mA Transcranial Direct Current Stimulation
Brief Title: 4 mA tDCS, Estrogen, and Leg Muscle Fatigability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Thorsten Rudroff, Assistant Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202005124
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Results first posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: Healthy
Keywords: transcranial direct current stimulation; muscle fatigue; brain stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Eumenorrheic Women (Experimental): Participants will have the anode (active electrode) placed over the brain area that controls their dominant leg and the cathode (return electrode) above the ipsilateral eyebrow. tDCS is administered in the early follicular phase, late follicular phase, and mid-luteal phase of their menstrual cycle.
  tDCS: Stimulation is ramped up to 4 mA over the first 30 seconds and stays at 4 mA for the remainder of the simulation time.
  Sham: Stimulation is turned on (4 mA) for 30 seconds at the beginning and the end of the trial but stays at 0 mA in the intervening time.
  Interventions: Device: Sham transcranial direct current stimulation 4 mA; Device: Transcranial direct current stimulation 4 mA

INTERVENTIONS:
Device: Sham transcranial direct current stimulation 4 mA — Uses weak electrical current (4 mA intensity) at the beginning and the end of a given stimulation period to control for potential placebo-like effects or participant expectation bias.
  Other Names: Sham tDCS 2 mA
Device: Transcranial direct current stimulation 4 mA — Uses weak electrical current (4 mA intensity) to either increase or decrease brain excitability and improve functional or cognitive outcomes.
  Other Names: tDCS 4 mA

SUMMARY:
The majority of transcranial direct current stimulation (tDCS) studies have failed to consider sex as a modulating factor. This neglect may partly account for the high inter-subject variability bemoaned by many tDCS investigators (e.g., approximately 50% of participants do not respond to tDCS) and has certainly delayed progress in the field. Therefore, research into how sex influences stimulation-related outcomes is vital to fully understand the underlying mechanisms of tDCS, which has shown great inconsistency.

Because of the menstrual cycle, the hormonal levels of women fluctuate considerably more than in men. Importantly, these hormonal variations might impact the efficacy of neuromodulatory tools, like tDCS. It is suggested that estrogen, which is high in the second follicular phase, reinforces excitatory mechanisms in the motor cortex. However, because anodal tDCS enhances cortical excitation there is also a possibility of excessive excitability. For instance, anodal tDCS may lead to overexcitation and non-optimal performance when it is applied in the second follicular phase of the menstrual cycle. Currently, there is a lack of knowledge on how the phases of the menstrual cycle affect tDCS performance outcomes in healthy young women because no studies have examined if and how the phases of the menstrual cycle alter tDCS efficacy.

This study is critical for determining the optimal time to administer anodal tDCS, and the ideal intensity for that administration, to achieve the most beneficial results. Furthermore, this investigation will emphasize the need for future tDCS studies to test women during the same menstrual cycle phase.

DETAILED DESCRIPTION:
The majority of transcranial direct current stimulation (tDCS) studies have failed to consider sex as a modulating factor. This neglect may partly account for the high inter-subject variability bemoaned by many tDCS investigators (e.g., approximately 50% of participants do not respond to tDCS) and has certainly delayed progress in the field. Therefore, research into how sex influences stimulation-related outcomes is vital to fully understand the underlying mechanisms of tDCS, which has shown great inconsistency.

Because of the menstrual cycle, the hormonal levels of women fluctuate considerably more than in men. There are two main phases of the menstrual cycle: 1) the follicular phase, characterized by low levels of estradiol and progesterone (first follicular phase, days 1-7) followed by increased levels of estradiol and low levels of progesterone (second follicular phase, days 7-14); and 2) the luteal phase (days 14-28), characterized by moderate estradiol and high progesterone levels. Importantly, these hormonal variations might impact the efficacy of neuromodulatory tools, like tDCS.

It is suggested that estrogen, which is high in the second follicular phase, reinforces excitatory mechanisms in the motor cortex. Thus, it appears that higher levels of estradiol increase cortical excitability. However, because anodal tDCS enhances cortical excitation there is also a possibility of excessive excitability. For instance, anodal tDCS may lead to overexcitation and nonoptimal performance when it is applied in the second follicular phase of the menstrual cycle. Currently, there is a lack of knowledge on how the phases of the menstrual cycle affect tDCS performance outcomes in healthy young women because no studies have examined if and how the phases of the menstrual cycle alter tDCS efficacy.

This research will be significant because the changing hormone levels during the different phases of menstruation in women is an especially important factor for minimizing response variability from tDCS. Thus, this study is critical for determining the optimal time to administer anodal tDCS, and the ideal intensity for that administration, to achieve the most beneficial results. Furthermore, this investigation will emphasize the need for future tDCS studies to test women during the same menstrual cycle phase.

ELIGIBILITY:
Inclusion Criteria:

1. Has a regular menstrual cycle
2. Young adult (18-35 years)
3. Right-side dominant
4. At least 30 min of moderate-intensity, physical activity on at least 3 days of the week for at least the last 3 months
5. Without chronic neurological, psychiatric, or medical conditions
6. Not taking any psychoactive medications.

Exclusion Criteria:

1. Pregnant
2. Known holes or fissures in the skull
3. Metallic objects or implanted devices in the skull (e.g., metal plate)
4. Women on hormonal contraceptives/supplements.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Rudroff, PhD, Principal Investigator — Health and Human Physiology
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eumenorrheic Women
Started | 10
tDCS, Early Follicular Phase | 10
Sham, Early Follicular Phase | 10
tDCS, Late Follicular Phase | 10
Sham, Late Follicular Phase | 10
tDCS, Mid-Luteal Phase | 10
Sham, Mid-Luteal Phase | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Eumenorrheic Women: Biological women will have the anode (active electrode) placed over the brain area the controls their dominant leg and the cathode (return electrode) above the eyebrow on the opposite side of the head.
  Transcranial direct current stimulation 2 mA: Uses weak electrical current (2 mA intensity) to either increase or decrease brain excitability and improve functional or cognitive outcomes. Stimulation is ramped up to 2 mA over the first 30 seconds and stays at 2 mA for the remainder of the stimulation time.
  Sham transcranial direct current stimulation 2 mA/4mA: Uses weak electrical current (2 mA or 4 mA intensity) at the beginning and the end of a given stimulation period to control for potential placebo-like effects or participant expectation bias. Stimulation is turned on (2 mA or 4 mA) for the 30 seconds at the beginning and the end of the trial but stays at 0 mA in the intervening time.
Arm/Group | Eumenorrheic Women
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Index From the Isokinetic Fatigue Test
Description: Perform 40 consecutive flexion and extension repetitions of the knee on the dominant leg. After a 10 minute rest, do the same task on the non-dominant leg.
  The fatigue index was calculated using the greatest torque from the relevant repetitions of the fatigue test as follows: ([mean of reps 3 through 7-mean of last five reps]/mean of reps 3 through 7) X 100 and is expressed as a percentage of decline in torque production.
Time Frame: Completed at each visit, spaced approximately 14 days apart for 2 consecutive months
Measure: Mean (Standard Deviation); unit: Percent decline
Arm/Group | Eumenorrheic Women
Number analyzed (Participants) | 10
Percent decline
  tDCS High Estrogen | 61.7 (10.6)
  Sham High Estrogen | 46.7 (20.0)
  tDCS Low Estrogen | 57.28 (11.57)
  Sham Low Estrogen | 55.90 (8.67)
Statistical Analysis 1: Comparison: Eumenorrheic Women; Test type: Superiority; p < 0.05, ANOVA — Post hoc analyses (paired t-tests and Bonferroni correction) and effect size (Cohen's d) were calculated to clarify significant main effects and interactions; Normality and sphericity evaluated with Shapiro-Wilk test and Mauchly's test. Greenhouse-Geisser corrections used when sphericity was violated

2. Primary Outcome: Muscle Activity During the Strength and Fatigue Tests
Description: Collect electromyographic (EMG; muscle activity) information during the fatigue tests. Muscle activity is measured as electrical signals/voltages.
  The muscle activity of the knee extensors (rectus femoris, vastus medialis, and vastus lateralis) was averaged to represent the cumulative activity of this muscle group. The first two repetitions of the fatigue test were considered adaptation repetitions and were removed. Therefore, the remaining 38 repetitions were used for the average EMG analyses. The subsequent 38 repetitions were also organized into 8 windows. The first seven windows consisted of five consecutive and non-overlapping repetitions (e.g., window 2 = reps 8-12; window 3 = reps 13-17, etc.) while the last (eighth) window was comprised of the final three repetitions.
Time Frame: Completed at each visit, spaced approximately 14 days apart for 2 consecutive months
Measure: Mean (Standard Deviation); unit: Microvolts
Arm/Group | Eumenorrheic Women
Number analyzed (Participants) | 10
Microvolts
  tDCS High Estrogen | 95.15 (26.46)
  tDCS Low Estrogen | 91.83 (16.48)
  Sham High Estrogen | 77.53 (19.71)
  Sham Low Estrogen | 82.35 (21.44)
Statistical Analysis 1: Comparison: Eumenorrheic Women; Test type: Superiority; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Estrogen Level
Description: Staff nurses collected 4.5 mL of blood from the median cubital vein of the left arm (total volume collected per subject = 9 mL) for the estrogen assay. Samples were immediately analyzed for serum estrogen levels after the blood draws by University of Iowa Hospitals and Clinics Pathology technicians using an Electrochemiluminescence Assay (Roche Diagnostics, Basel, Switzerland). The estrogen assay had a lower limit of detection of 5 pg/mL and a coefficient of variation of 8%.
  Because menstrual cycles have great inter- and intrasubject variability, the peak estrogen levels of the subjects were not consistently found in the late-follicular phase, which is a common failing of menstrual cycle phase calendar estimation. Thus, estrogen levels were grouped as high or low according to each individual subject's estrogen serum levels, irrespective of the anticipated/targeted phase.
Time Frame: Completed at each visit, spaced approximately 14 days apart for 2 consecutive months
Measure: Mean (Standard Deviation); unit: (pg/mL)
Arm/Group | Eumenorrheic Women
Number analyzed (Participants) | 10
(pg/mL)
  tDCS High Estrogen | 157.7 (101.5)
  tDCS Low Estrogen | 31.9 (10.9)
  Sham High Estrogen | 137.2 (114.0)
  Sham Low Estrogen | 42.9 (25.1)

ADVERSE EVENTS:
Time Frame: Completed at each visit, spaced approximately 14 days apart for 2 consecutive months
Description: This study was deemed to be of non-significant risk. This type of brain stimulation has established safety and tolerability data in both human and animal models.
Arm/Group | Eumenorrheic Women
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT04471805/Prot_SAP_001.pdf